CLINICAL TRIAL: NCT00686348
Title: Somatuline® Depot (Lanreotide) Injection for Acromegaly (SODA): A Post-marketing Observational Study
Brief Title: Somatuline® Depot (Lanreotide) for Acromegaly Post-Marketing Observational Study
Acronym: SODA
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-TL-52030-225 (MS319)
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
Keywords: acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Routine clinical laboratory assessments will be performed: GH and IGF-1
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the safety and effectiveness of Somatuline® Depot (lanreotide) Injection when administered by a health care professional (HCP), the patient, the patient's partner or parent/guardian as part of their routine acromegaly care.

DETAILED DESCRIPTION:
The objectives of this post-marketing observational study are to assess the safety and effectiveness, as measured by insulin-like growth factor-1 (IGF-1) and growth hormone (GH) levels, of Somatuline® Depot (lanreotide) Injection when administered by a health care professional (HCP), the patient, the patient's partner or parent/guardian as part of their routine acromegaly care. Treatment convenience and acromegaly symptom relief will also be assessed through questionnaires, and demographic and medical history information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a clinical diagnosis of acromegaly
* The patient must be treated with Somatuline® Depot (including patients newly prescribed Somatuline® Depot)
* The patient or legally authorized representative must be able to understand the protocol and give signed informed consent. Assent from the patient should also be obtained, where appropriate. Signed informed consent and assent must be obtained before any study-related activities are conducted.

Exclusion Criteria:

* Symptomatic, untreated biliary lithiasis
* Known hypersensitivity to somatostatin analogs or related compounds (e.g., octreotide)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a clinical diagnosis of acromegaly
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2008-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Assess the safety & effectiveness, as measured by IGF-1 & GH levels, of Somatuline® Depot Injection when administered by a health care professional, the patient, the patient's partner or parent/guardian as part of their routine acromegaly care. | 2 - 4 years/patient

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen (formerly Tercica, Inc.)
Locations (1):
- Ipsen, Basking Ridge, New Jersey, United States

REFERENCES:
- [Derived] Salvatori R, Gordon MB, Woodmansee WW, Ioachimescu AG, Carver DW, Mirakhur B, Cox D, Molitch ME. A multicenter, observational study of lanreotide depot/autogel (LAN) in patients with acromegaly in the United States: 2-year experience from the SODA registry. Pituitary. 2017 Dec;20(6):605-618. doi: 10.1007/s11102-017-0821-y. PMID 28741071
- See also: Tercica Somatuline Depot General Information — http://www.somatulinedepot.com/